CLINICAL TRIAL: NCT00001023
Title: Evaluation of the Safety, Tolerance and Pharmacokinetics of Rifabutin/Clarithromycin Combination and Rifabutin/Azithromycin Combination in HIV-Infected Patients
Brief Title: The Safety and Effectiveness of Rifabutin, Combined With Clarithromycin or Azithromycin, in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DATRI 001; 11732 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Drug Interactions; Azithromycin; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections | interventions — Clarithromycin; Azithromycin; Rifabutin

INTERVENTIONS:
Drug: Clarithromycin
Drug: Azithromycin
Drug: Rifabutin

SUMMARY:
PER 03/10/94 AMENDMENT: PART B. To determine whether there is an effect on plasma drug levels of azithromycin and rifabutin as measured by changes in the plasma concentration-time curve (AUC) when these drugs are taken concomitantly.

ORIGINAL PRIMARY: To gain preliminary information about the safety and tolerance of clarithromycin and azithromycin in combination with rifabutin (three potential agents against Mycobacterium avium-intracellulare) in HIV-infected patients with CD4 counts < 200 cells/mm3.

ORIGINAL SECONDARY: To determine whether there is an effect on the pharmacokinetics of the macrolide antibiotics or rifabutin when these drugs are taken concomitantly. To monitor the effect of rifabutin therapy on dapsone serum levels in patients taking dapsone for PCP prophylaxis. To monitor the effect of macrolide/rifabutin combination therapies on AZT or ddI serum levels.

Two new macrolide antibiotics, clarithromycin and azithromycin, and rifabutin (a rifamycin derivative) have all demonstrated in vitro and in vivo activity against Mycobacterium avium-intracellulare, a common systemic bacterial infection complicating AIDS. Further information is needed, however, regarding the clinical and pharmacokinetic interaction of these drugs used in combination.

DETAILED DESCRIPTION:
Two new macrolide antibiotics, clarithromycin and azithromycin, and rifabutin (a rifamycin derivative) have all demonstrated in vitro and in vivo activity against Mycobacterium avium-intracellulare, a common systemic bacterial infection complicating AIDS. Further information is needed, however, regarding the clinical and pharmacokinetic interaction of these drugs used in combination.

AMENDED 03/10/94 (Part B): Approximately 38 HIV-infected or uninfected subjects are randomized to receive azithromycin or rifabutin (Groups 3 and 4) daily for 14 days, followed by a combination regimen of both drugs for 4 additional weeks. Patients are followed weekly. Pharmacokinetic sampling will be performed on days 14, 15, and 42-45.

ORIGINAL: Sixty-eight patients are randomly assigned to one of four groups (17 patients per group). They receive either clarithromycin or azithromycin in combination with rifabutin on one of two different dosing schedules. Patients receive medication for 6 weeks and undergo follow-up weekly during drug administration and at week 8.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Primary or secondary PCP prophylaxis with TMP/SMX, dapsone, or aerosolized pentamidine.
* Any approved therapy for antiretroviral treatment, or antiretroviral therapy available through FDA-sanctioned treatment IND or treatment protocol.

Patients must have:

AMENDED (PART B):

* Either HIV infection OR no HIV infection.
* CD4 count unspecified.

ORIGINAL:

* Documented HIV infection.
* CD4 count < 200 cells/mm3 within 90 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known Mycobacterium avium-intracellulare (MAI) bacteremia or presence of a clinical syndrome compatible with MAI (i.e., fevers, weight loss, elevated LDH and alkaline phosphatase).
* Fever = or > 38.5 deg C (100.4 deg F) within 7 days prior to study entry.

Concurrent Medication:

Excluded:

* Acute or chronic use of phenobarbital, carbamazepine, rifampin, dilantin, fluconazole, itraconazole, ketoconazole, ciprofloxacin, beta-blockers, or clarithromycin.
* Oral contraceptives.
* Acute therapy for an AIDS-related opportunistic infection or malignancy, or other acute medical illness, or infection.
* Maintenance therapy for CMV, cryptococcal meningitis, or toxoplasmosis.
* Cytotoxic chemotherapy.

Patients with the following prior conditions are excluded:

* History of intolerance or hypersensitivity to study drugs, other macrolide antibiotics, or rifampin.
* Three or more loose bowel movements per day within 3 months prior to study entry.
* Unintentional weight loss >= 5 percent of body weight within 3 months prior to study entry.

Prior Medication:

Excluded:

* Rifabutin within 30 days prior to study entry.
* Clarithromycin or azithromycin within 14 days prior to study entry.
* Acute therapy for an AIDS-related opportunistic infection or malignancy, or other acute medical illness, or infection within 28 days prior to study entry.

Prior Treatment:

Excluded:

* Blood transfusions within 1 month prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Hafner, Study Chair; H Standiford, Study Chair
Locations (11):
- United States (11):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - Davies Med Ctr, San Francisco, California
  - Denver Public Health Dept, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Tulane Univ Med School, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Veterans Adm, Baltimore, Maryland
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Univ of Rhode Island / Roger Williams Med Ctr, Providence, Rhode Island
  - Med College of Virginia / School of Pharmacy, Richmond, Virginia

REFERENCES:
- [Background] Hafner R, Bethel J, Standiford HC, Follansbee S, Cohn DL, Polk RE, Mole L, Raasch R, Kumar P, Mushatt D, Drusano G; DATRI 001B Study Group. Tolerance and pharmacokinetic interactions of rifabutin and azithromycin. Antimicrob Agents Chemother. 2001 May;45(5):1572-7. doi: 10.1128/AAC.45.5.1572-1577.2001. PMID 11302832